CLINICAL TRIAL: NCT04986969
Title: Online Cognitive Behavioral Therapy for Depressive Symptoms in Rural Patients with Coronary Heart Disease
Brief Title: Online Cognitive Behavioral Therapy for Depressive Symptoms in Rural Patients with Cardiac Disease
Acronym: COMBAT-DS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Debra Moser (Other)
Collaborators: University of California, Los Angeles (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor-Investigator, Debra Moser, Professor and Linda C Gill Endowed Chair of Nursing, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AD-2019C3-17982
Record Dates: First submitted 2021-07-13; First posted 2021-08-03 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Depressive Symptoms; Heart Diseases
Keywords: rural; cardiac diseases; depressive symptoms; cognitive behavioral therapy
MeSH Terms: conditions — Depression; Heart Diseases

STUDY DESIGN:
Intervention Model Description: The investigators will use a longitudinal, 2-arm randomized, comparative effectiveness trial, stratified by sex. Patients will be randomized to one of two study arms: 1) real-time, face-to-face, video-conferenced CBT (vcCBT) with a trained CBT therapist; or 2) self-administered internet-based CBT (iCBT) via a well-tested online CBT program, MoodGym. Patients will be followed for 12 months from baseline and depressive symptom data collected at 3, 6, and 12 months to characterize intervention response. Participants will be randomized to either vcCBT (n = 150) or iCBT (n = 150) arm.
Who Masked: Investigator
Masking Description: Active therapy is delivered to patients, thus it is impossible to mask the participant or care provider. The investigators are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- real-time, face-to-face, video-conferenced CBT (vcCBT) (Active Comparator): vcCBT is cognitive behavioral therapy that consists of eight face-to-face video-conferencing sessions via tablet computers lasting approximately 45 minutes each.
  Interventions: Behavioral: Online cognitive behavioral therapy
- self-administered internet-based CBT (iCBT) (Active Comparator): iCBT is self-directed cognitive behavioral therapy using an interactive internet program, MoodGYM, which does not include direct interactions with a therapist.
  Interventions: Behavioral: Online cognitive behavioral therapy

INTERVENTIONS:
Behavioral: Online cognitive behavioral therapy — online cognitive behavioral therapy delivered using one of two active methods

SUMMARY:
Individuals with heart disease and depressive symptoms suffer from higher death rates, higher rates of acute cardiac events (such as heart attacks), and faster progression of heart disease compared to those with heart disease who do not have depressive symptoms, and these problems are much worse in rural people. Unfortunately, rural people with heart disease and depressive symptoms do not receive needed therapy for depressive symptoms because of lack of mental health providers in rural areas, worries about stigma, and difficulty accessing mental health care because of multiple barriers to traveling to get care. To overcome these barriers, the investigators will compare the impact of two types of online cognitive behavioral therapy (video-conferenced face-to-face versus self-administered internet-based) and usual care on depressive symptoms to provide patients and healthcare providers with needed information about which is more effective and to increase the number of patients adequately treated.

DETAILED DESCRIPTION:
Rural areas are noted for marked disparities in mortality, cardiovascular health, and access to health care. Prevalence rates for both coronary heart disease (CHD) and depressive symptoms in rural areas are higher than in urban areas. These facts are important because CHD patients experience high rates of depressive symptoms, which are associated with increased risk of getting and dying from CHD. Unfortunately, rural people with CHD and depressive symptoms do not receive needed therapy for depressive symptoms because of lack of mental health providers in rural areas, worries about stigma leading to treatment avoidance, and difficulty accessing mental health care because of barriers to travel to get care. Cognitive behavioral therapy (CBT), reduces depressive symptoms in CHD patients, but in its traditional form (in-person meetings of patient and therapist), CBT is resource-intensive and inaccessible to most rural patients. Wireless internet technology has the potential to make CBT more user-friendly, and accessible to rural patients. There has been a proliferation of alternative, internet-based, remote-delivery CBT interventions recently. The permutations of remote-delivery CBT fall under two categories - real-time, face-to-face, video-conferenced CBT (vcCBT) and self-administered internet-based CBT (iCBT). It is unclear which category of these delivery modalities is more effective. Determining which treatment option is more effective for treating depressive symptoms in rural patients with CHD and depressive symptoms will identify an easily accessible treatment option for rural patients. Using a randomized, controlled, stratified (by sex) design, the investigators will compare vcCBT, iCBT and usual care in rural CHD patients on the primary outcome of depressive symptoms over time. In addition, the investigators will determine whether intervention adherence, satisfaction or acceptability moderate treatment effects. The investigators will also assess whether sex or stigma moderate intervention effects to determine whether effectiveness of treatment option varies by sex or stigma level. Data about outcomes will be collected at baseline, 3 months, 6 months, and 12 months and provide important information about the trajectory of outcomes. Results from this study will provide new knowledge about which approach to treating depressive symptoms in rural CHD patients is more effective to improve decision-making in patients and healthcare providers, and increase the number of patients properly treated.

ELIGIBILITY:
Inclusion Criteria:

* at least moderate depressive symptoms (PHQ-9 ≥ 10)
* rural dwelling
* has had physician-documented acute coronary syndrome (ACS) event

Exclusion Criteria:

* cognitive impairment
* major psychiatric comorbidities, which might require additional treatment
* presence of non-CHD conditions likely to be fatal within next year.

Ages: 21 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms as a result of intervention effects | Baseline, 3, 6 and 12 months
  Change in levels of depressive symptoms measured using the Patient Health Questionnaire-9, across time and between subjects. The Patient Health Questionnaire-9 is a measure that consists of nine items that correspond to criteria for diagnosing depression. Higher scores indicate greater severity of symptoms. Scores on measure can range from 0-27 with an accepted cut-off of ≥ 10 for moderate symptoms. Reliability and validity of the instrument have been established in a variety of populations, including cardiac patients.
Change in intervention effects on depressive symptoms moderated by perceived stigma | Baseline, 3, 6, and 12 months
  The investigators will determine whether perceived stigma moderates intervention effects on depressive symptoms across time. Stigma refers to negative beliefs about a condition and its treatment. Depression-related stigma will be measured using the Depression Stigma Scale. Developed to measure personal stigma related to being treated for depressive symptoms, the measure has been used extensively since its inception. Scores on the 18-item total scale can range from 0-36, and higher scores indicate greater perceptions of stigma. The instrument has well-established reliability and validity, and has been used in rural Kentuckians.
Change in intervention effects on depressive symptoms moderated by sex | Baseline, 3, 6, and 12 months
  The investigators will determine whether sex moderates intervention effects on depressive symptoms across time. Sex will be self-described by the patient.

SECONDARY OUTCOMES:
Change in intervention effects on depressive symptoms moderated by health literacy | Baseline, 3, 6, and 12 months
  Determine whether health literacy measured using the Newest Vital Sign moderates intervention effects on change in depressive symptoms. Health literacy is defined as the degree to which individuals have the capacity to obtain, process, and understand basic health information and services needed to make appropriate health decisions. The investigator will assess health literacy using the Newest Vital Sign. This instrument is sensitive, reliable and valid for the assessment of health literacy, and is well-accepted by individuals being screened even when they have low educational level.
Compare all-cause hospitalization rates between intervention groups | 3 months
  Measurement of hospitalization rates using the electronic health record and patient interview
Compare all-cause hospitalization rates between intervention groups | 6 months
  Measurement of hospitalization rates using the electronic health record and patient interview
Compare all-cause hospitalization rates between intervention groups | 12 months
  Measurement of hospitalization rates using the electronic health record and patient interview
Compare physical activity levels between groups | 3 months
  Measurement of physical activity levels using actigraphy. Actigraphy is an objective method of obtaining accurate and reproducible activity levels, and advances in the technology have produced an instrument that reliably and validly represents physical activity levels. The investigators use the GT9X-BT Link Bluetooth Activity Monitor (ActiGraph, Pensacola, FL). The Actigraph is an omni-directional accelerometer, which assesses acceleration in multiple directions as opposed to uniaxial accelerometer, which is sensitive to movement only in the vertical axis. The actigraph has a dynamic range of ± 8 g. The Actigraph allows researchers to estimate energy expenditure by quantifying the amount time spent in light [<3 metabolic equivalents (METs)], moderate (3-5.99 METs), and vigorous (≥6 METs) physical activity.
Compare physical activity levels between groups | 6 months
  Measurement of physical activity levels using actigraphy. Actigraphy is an objective method of obtaining accurate and reproducible activity levels, and advances in the technology have produced an instrument that reliably and validly represents physical activity levels. The investigators use the GT9X-BT Link Bluetooth Activity Monitor (ActiGraph, Pensacola, FL). The Actigraph is an omni-directional accelerometer, which assesses acceleration in multiple directions as opposed to uniaxial accelerometer, which is sensitive to movement only in the vertical axis. The actigraph has a dynamic range of ± 8 g. The Actigraph allows researchers to estimate energy expenditure by quantifying the amount time spent in light [<3 metabolic equivalents (METs)], moderate (3-5.99 METs), and vigorous (≥6 METs) physical activity.
Compare physical activity levels between groups | 12 months
  Measurement of physical activity levels using actigraphy. Actigraphy is an objective method of obtaining accurate and reproducible activity levels, and advances in the technology have produced an instrument that reliably and validly represents physical activity levels. The investigators use the GT9X-BT Link Bluetooth Activity Monitor (ActiGraph, Pensacola, FL). The Actigraph is an omni-directional accelerometer, which assesses acceleration in multiple directions as opposed to uniaxial accelerometer, which is sensitive to movement only in the vertical axis. The actigraph has a dynamic range of ± 8 g. The Actigraph allows researchers to estimate energy expenditure by quantifying the amount time spent in light [<3 metabolic equivalents (METs)], moderate (3-5.99 METs), and vigorous (≥6 METs) physical activity.
Compare medication adherence between groups | 3 months
  Measurement of medication adherence will be done using the Medication Event Monitoring System. Medication adherence will be measured with the Medication Event Monitoring System (MEMS; AARDEX, Union City, CA), a reliable, accurate and objective method. The MEMS is considered the gold standard in medication adherence measurement. The MEMS offers the advantage of objective measurement and has been successfully used in multiple clinical trials by our group.
Compare medication adherence between groups | 6 months
  Measurement of medication adherence will be done using the Medication Event Monitoring System. Medication adherence will be measured with the Medication Event Monitoring System (MEMS; AARDEX, Union City, CA), a reliable, accurate and objective method. The MEMS is considered the gold standard in medication adherence measurement. The MEMS offers the advantage of objective measurement and has been successfully used in multiple clinical trials by our group.
Compare medication adherence between groups | 12 months
  Measurement of medication adherence will be done using the Medication Event Monitoring System. Medication adherence will be measured with the Medication Event Monitoring System (MEMS; AARDEX, Union City, CA), a reliable, accurate and objective method. The MEMS is considered the gold standard in medication adherence measurement. The MEMS offers the advantage of objective measurement and has been successfully used in multiple clinical trials by our group.
Compare the effect of intervention effects on within-meal, across meal, and within-food group diet variety | Baseline
  Measured using interviews for dietary recall
Compare the effect of intervention effects on within-meal, across meal, and within-food group diet variety | 3 months
  Measured using interviews for dietary recall
Compare the effect of intervention effects on within-meal, across meal, and within-food group diet variety | 6 months
  Measured using interviews for dietary recall
Compare the effect of intervention effects on within-meal, across meal, and within-food group diet variety | 12 months
  Measured using interviews for dietary recall

CONTACTS AND LOCATIONS:
Overall Officials: Debra K Moser, PhD, RN, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
We will use the PCORI-prescribed methods for data-sharing. Deidentified data including the major primary outcome data will be made available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available 12 months after the end of the study. It will be available in the University of Michigan data repository (per PCORI) forever.
Access Criteria: Request from the repository.

REFERENCES:
- [Derived] Tully PJ, Ang SY, Lee EJ, Bendig E, Bauereiss N, Bengel J, Baumeister H. Psychological and pharmacological interventions for depression in patients with coronary artery disease. Cochrane Database Syst Rev. 2021 Dec 15;12(12):CD008012. doi: 10.1002/14651858.CD008012.pub4. PMID 34910821